CLINICAL TRIAL: NCT03999229
Title: Phase 1 Study of S-Nitrosylation Therapy to Improve Tissue Oxygenation During Autologous Blood Transfusion in Healthy Volunteer
Brief Title: S-Nitrosylation (SNO) Therapy During Autologous Blood Transfusion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: James Reynolds (Other)
Collaborators: Case Western Reserve University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, James Reynolds, Professor of Anesthesiology and Perioperative Medicine and a member of the Case Institute for Transformative Molecular Medicine, Case Western Reserve University
Organization: Case Western Reserve University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20221492; 5R01HL126900 (NIH)
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Transfusion Related Complication
Keywords: S-Nitrosylation; Tissue Oxygenation; Anemia-induced tissue hypoxia; Red blood cell Transfusion
MeSH Terms: interventions — Saline Solution; Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: This is an open-label phase I trial. Healthy young adult volunteers that would considered eligible by American Red Cross standards to donate blood will be screened by qualified practitioners for eligibility to participate in the above mentioned study. We anticipate an accrual number of 35, with subjects randomized to receive their blood (n=30) or saline (n=5) while breathing an SNO agent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Blood transfusion with SNO agent (Active Comparator): Autologous blood transfusion packed red blood cells (RBCs) while inhaling S-nitrosylating agent (SNO)
  A single intra venous blood transfusion of one unit of packed Red Blood Cells (RBCs) will be given over the standard transfusion flow rate of 5 ml/min under the direction of a physician or a licensed medical professional.
  Inhalation of SNO agent, 20-40 parts per million will occur during the transfusion.
  Interventions: Drug: SNO; Drug: Red Blood Cell
- Normal Saline with SNO agent (Placebo Comparator): Normal Saline Transfusion while inhaling S-nitrosylating agent (SNO)
  A single intra venous infusion of one unit of normal saline, will be given over the standard transfusion flow rate of 5 ml/min under the direction of a physician or a licensed medical professional.
  Inhalation of the SNO agent at 40 parts per million, will occur during the transfusion.
  Interventions: Drug: SNO; Drug: Normal Saline

INTERVENTIONS:
Drug: SNO — S-nitrosylating agent (SNO) Inhalation
Drug: Normal Saline — Normal Saline transfusion
  Arms: Normal Saline with SNO agent
Drug: Red Blood Cell — Blood transfusion (RBCs)
  Arms: Blood transfusion with SNO agent

SUMMARY:
The Purpose of the study is to test the hypothesis that administration of an S-nitrosylating (SNO) agent can improve tissue oxygenation during transfusion of packed red blood cells (RBCs).

DETAILED DESCRIPTION:
Transfusion is the most common therapeutic intervention employed to maintain and/or improve tissue and end-organ oxygen delivery. Despite the conceptual simplicity of this treatment recent studies indicate that RBC infusion often produces little clinical benefit and may actually harm the recipient by exacerbating rather than correcting anemia-induced tissue hypoxia.

The main driver/regulator of tissue oxygenation is blood flow not blood oxygen content. In turn flow into the microvasculature is controlled by small molecules called S-nitrosothiols (SNOs), the most important of which is S-nitrosylated hemoglobin (SNO-Hb).

The investigators determined that storage of human blood leads to rapid losses in SNO-Hb that are precisely paralleled by losses in the ability of stored RBCs to dilate blood vessels and thereby deliver oxygen. The investigators have now recently completed an autologous human blood transfusion that confirms the pre-clinical findings in that administration of 1 unit of packed RBCs to young healthy subjects did not improve tissue oxygenation and reduced circulating SNO-Hb levels.

This novel mechanism for the loss of physiological activity in banked blood and, more importantly, a putative intervention for its correction, raise the possibility that restoration of NO bioactivity could correct the deficit in oxygen delivery. As such, The Investigators plan to repeat our transfusion study with the addition of administering an S-nitrosylating agent during RBC infusion.

ELIGIBILITY:
Eligibility Criteria

Recruiting and studying of healthy human subjects with no pre-existing pathologic conditions from the local population. As a result the inclusion criteria is deliberately broad.

Inclusion Criteria

1. Hemoglobin > 12 g/dl
2. Healthy, non-pregnant adults with no pre-existing blood disorders or disease states that impact oxygen delivery.

2a. Active blood and platelet donors will be sought as study participants since these individuals are familiar with the routines for blood withdrawal and re-infusion.

Exclusion Criteria

The exclusion criteria is derived from the American Red Cross(ARC) Standard Operating Procedure (SOP) for autologous donation AND the parameters set out in the investigational new drug application (IND).

1. Individuals who are pregnant, breastfeeding, or are unwilling to avoid pregnancy during the study.
2. Individuals with an anatomic anomaly that would increase the risks associated with placement of the vascular catheters.
3. Individuals who report chronic diseases requiring medication of the heart, lungs, kidney, liver, etc or afflicted with any acute or chronic pathology that in the opinion of the screening physician makes them unsuitable for study.
4. Individuals with a recent history of antibiotic therapy (check for underlying cause).
5. Individuals unwilling to refrain from taking any phosphodiesterase 5 (PDE-5) inhibitor for at least 24 h prior to donation and/or autologous transfusion.
6. Individuals taking a vitamin K antagonist (warfarin) or other anticoagulant (e.g. heparin, clopidogrel, enoxaparin or dalteparin).
7. Individuals taking allopurinol, beta-adrenergic blockers, tricyclic antidepressants, meperidine (or related central nervous system (CNS) agents), or nitrates.
8. Individuals on long-term antihistamine therapy 8a. The study physician will determine on a case by case basis the suitability for inclusion of individuals who control seasonal or acute allergies with occasional antihistamine use.
9. Individuals with blood pressure parameters outside the normal range, i.e., higher than 130 mm Hg systolic and/or higher than 90 mm Hg diastolic; mild hypertension is acceptable by the Red Cross for blood donation.
10. Individuals with heart rates outside the range of 50 to 100 beats per minutes or with a pathologic irregularity.

10a. Pulses lower than 50 may be acceptable if the study participant participates in endurance training. The study physician will be consulted for evaluation.

11. Individuals with an inherited or acquired blood coagulation disorder, congenital methemoglobinemia, or a familial hemoglobinopathy that impacts oxygen delivery (e.g. sickle cell).

12. Individuals with any illness that may increase the risks associated with the study.

13. Individuals who previously received blood products to treat an acute condition will be evaluated on a case by case basis.

14. Individuals who report an acute or chronic disease state that may impact oxygen delivery.

15. Individuals with evidence of diminished lung capacity.

16. Individuals who might have difficulty with the placement of a face mask (e.g. claustrophobia, uncontrolled asthma, severe allergies, sensitive skin) and/or the inhalation of a product for approximately 2-3 hours.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Peripheral Tissue Oxygenation | Monitoring is continuous once the probes are placed on the skin. It will start approximately 30 minutes prior to blood transfsuion and continue overnight and then stopped next morning when subject is discharged. Total time is up to 24 hours.
  Measurement of small vessel blood flow and oxygenation status with near infrared spectroscopy (NIRS).
  NIRS can record the amount of oxygenated and de-oxygenated hemoglobin (the main protein in red blood cells) using different light frequencies shined through probes attached to the skin. The tissue oxygenation measurement is expressed as a percentage based on the ratio of oxygenated to de-oxygenated hemoglobin. It is continually-measured to see if it is changing in response to transfusion or administration of the study drug.
Oxygen Utilization | Blood samples are obtained every 3 to 6 hours before during and after blood transfsuion until subject is discharged Total time is up to 24 hour
  Determined by measuring arterial and venous blood oxygen levels - Blood Gas (BG)
  A BG is a test that measures the the levels of oxygen (O2) in the blood obtained from an artery or vein. The test is used to check the function of the patient's lungs and how well they are able to move oxygen around the body.
  The amount of oxygen is expressed as percent of the overall amount of hemoglobin. The difference in the amount of oxygen in arterial and venous blood is calculated as the measure of oxygen utilization and if it is changing in response to transfusion or administration of the study drug.

SECONDARY OUTCOMES:
Kidney Function Test | Blood samples are obtained every 3 to 6 hours before during and after blood transfsuion until subject is discharged Total time is up to 24 hour
  Blood samples will be assayed for markers of kidney function:
  creatinine - milligram per deciliter
  albumin - grams per deciliter
  blood urea nitrogen - milligram per deciliter
  This 3 blood markers are incorporated into a formula to calculate glomerular filtration rate or GFR. This is a measure of how well your kidneys are filtering your blood and if it is changing in response to transfusion or administration of the study drug.
Liver Function Test | Blood samples are obtained every 3 to 6 hours before during and after blood transfsuion until subject is discharged Total time is up to 24 hour
  Blood samples will be assayed for markers of liver function:
  alanine transaminase or ALT - units per liter
  aspartate aminotransferase or AST - units per liter
  The individual values are determined then the AST/ALT ratio is calculated to provide further information on liver status and if it is changing in response to transfusion or administration of the study drug.
Assessment of Immune Status | Blood samples are obtained every 3 to 6 hours before during and after blood transfsuion until subject is discharged Total time is up to 24 hour
  The number of white blood cells is counted in each blood sample. White blood cells (also called leukocytes) are an important measure of how the immune system is working and if it is changing in response to transfusion or administration of the study drug.
  leukocytes - reported as cell counts

CONTACTS AND LOCATIONS:
Overall Officials: James D. Reynolds, PhD, Principal Investigator — Case Western Reserve University; Mada Helou, MD, Study Director — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification and analysis will be shared.
Supporting Information: SAP, CSR
Time Frame: Available Immediately following publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Reynolds JD, Ahearn GS, Angelo M, Zhang J, Cobb F, Stamler JS. S-nitrosohemoglobin deficiency: a mechanism for loss of physiological activity in banked blood. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17058-62. doi: 10.1073/pnas.0707958104. Epub 2007 Oct 11. PMID 17940022
- [Background] Singel DJ, Stamler JS. Chemical physiology of blood flow regulation by red blood cells: the role of nitric oxide and S-nitrosohemoglobin. Annu Rev Physiol. 2005;67:99-145. doi: 10.1146/annurev.physiol.67.060603.090918. PMID 15709954
- [Background] McMahon TJ, Ahearn GS, Moya MP, Gow AJ, Huang YC, Luchsinger BP, Nudelman R, Yan Y, Krichman AD, Bashore TM, Califf RM, Singel DJ, Piantadosi CA, Tapson VF, Stamler JS. A nitric oxide processing defect of red blood cells created by hypoxia: deficiency of S-nitrosohemoglobin in pulmonary hypertension. Proc Natl Acad Sci U S A. 2005 Oct 11;102(41):14801-6. doi: 10.1073/pnas.0506957102. Epub 2005 Oct 3. PMID 16203976
- [Background] Pawloski JR, Hess DT, Stamler JS. Export by red blood cells of nitric oxide bioactivity. Nature. 2001 Feb 1;409(6820):622-6. doi: 10.1038/35054560. PMID 11214321
- [Background] VALTIS DJ. Defective gas-transport function of stored red blood-cells. Lancet. 1954 Jan 16;266(6803):119-24. doi: 10.1016/s0140-6736(54)90978-2. No abstract available. PMID 13118742
- [Background] Bunn HF, May MH, Kocholaty WF, Shields CE. Hemoglobin function in stored blood. J Clin Invest. 1969 Feb;48(2):311-21. doi: 10.1172/JCI105987. PMID 5764013
- [Background] Sugerman HJ, Davidson DT, Vibul S, Delivoria-Papadopoulos M, Miller LD, Oski FA. The basis of defective oxygen delivery from stored blood. Surg Gynecol Obstet. 1970 Oct;131(4):733-41. No abstract available. PMID 5458535
- [Background] Shah DM, Gottlieb ME, Rahm RL, Stratton HH, Barie PS, Paloski WH, Newell JC. Failure of red blood cell transfusion to increase oxygen transport or mixed venous PO2 in injured patients. J Trauma. 1982 Sep;22(9):741-6. doi: 10.1097/00005373-198209000-00004. PMID 7120526
- [Background] Rao SV, Jollis JG, Harrington RA, Granger CB, Newby LK, Armstrong PW, Moliterno DJ, Lindblad L, Pieper K, Topol EJ, Stamler JS, Califf RM. Relationship of blood transfusion and clinical outcomes in patients with acute coronary syndromes. JAMA. 2004 Oct 6;292(13):1555-62. doi: 10.1001/jama.292.13.1555. PMID 15467057
- [Background] Vincent JL, Baron JF, Reinhart K, Gattinoni L, Thijs L, Webb A, Meier-Hellmann A, Nollet G, Peres-Bota D; ABC (Anemia and Blood Transfusion in Critical Care) Investigators. Anemia and blood transfusion in critically ill patients. JAMA. 2002 Sep 25;288(12):1499-507. doi: 10.1001/jama.288.12.1499. PMID 12243637
- [Background] Malone DL, Dunne J, Tracy JK, Putnam AT, Scalea TM, Napolitano LM. Blood transfusion, independent of shock severity, is associated with worse outcome in trauma. J Trauma. 2003 May;54(5):898-905; discussion 905-7. doi: 10.1097/01.TA.0000060261.10597.5C. PMID 12777902